CLINICAL TRIAL: NCT06363669
Title: Acute Effects of Multi-ingredient Pre-workout Dietary Supplement on Physical Performance in Untrained Men
Brief Title: Effects of Caffeine-based Supplement on Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1_CAF_AWF
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Muscle Power
Keywords: exercise; caffeine; muscle power
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Group with placebo treatment (100 ml of orange-flavored water without any additional substances (0 kcal))
- group with MIPS supplementation (Experimental): Group with supplementation. Supplement was commercially available and dispensed without a prescription. The dietary supplement contained in one dose (30ml): beta-alanine 3000 mg, taurine 1000 mg, caffeine 290 mg, L-tyrosine 125 mg, and cayenne pepper extract (Capsicum annuum L.) 4.2 mg (of which 8% capsaicin). The supplement was mixed with water; in total, participants were given 100 ml of liquid to drink, 30 minutes before the warm-up for the all-out anaerobic test.
  Interventions: Dietary Supplement: multi-ingredient pre-workout dietary supplement (caffeine-based)

INTERVENTIONS:
Dietary Supplement: multi-ingredient pre-workout dietary supplement (caffeine-based) — The participants performed the exercise twice, in random order: as a control test and after supplement administration. The acute effects of MIPS supplementation (beta-alanine 3000 mg, taurine 1000 mg, caffeine 290 mg, L-tyrosine 125 mg, and cayenne pepper extract (Capsicum annuum L.) 4.2 mg (of which 8% capsaicin)) on aerobic and anaerobic performance were evaluated in untrained men
  Arms: group with MIPS supplementation

SUMMARY:
The aim of the study was to determine the acute effects of multi-ingredient pre-workout supple-ment (MIPS) containing: beta-alanine, taurine, caffeine, L-tyrosine, and cayenne pepper (capsaicin) on physical performance in untrained men

DETAILED DESCRIPTION:
The aim of our study was to determine the acute effects of commercially available multi-ingredient pre-workout supple-ment (MIPS) containing: beta-alanine, taurine, caffeine, L-tyrosine, and cayenne pepper (capsai-cin) on physical performance in untrained men. The aerobic and anaerobic capacity was determined after ingestion of MIPS. A randomized, crossover, single-blind design was used to evaluate the effects of the dietary supplement on physical performance. The participants performed the exercise test twice, in random order: as a control test and after supplement administration (MIPS). The measurements took place over two consecutive days. Somatic measurements were taken on the same day that the first all-out test was performed. Twelve young healthy men, without medical contraindications to supramaximal and maximal intensity exercise, participated in the study. The exercise tests took place under medical supervision.

ELIGIBILITY:
Inclusion Criteria:

lack of neuromuscular and musculoskeletal disorders; no medication nor dietary supplements used within the previous month which could potentially affect the study outcomes and self-described good health status. An additional inclusion criterion was the small amount of caffeine consumed per day, i.e. only one caffeinated coffee drink per day or less.

Exclusion Criteria:

consumption of energy drinks

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
anaerobic power | one day every 30 minutes
  Anaerobic power (anaerobic capacity) was determined twice (pre and post) dietary supplementation on one day. The anaerobic test was performed before supplemenation and 30 minutes after.
aerobic power | one day every 30 minutes
  Aerobic power (aerobic capacity) was determined twice (pre and post) dietary supplementation on one day. The anaerobic test was performed before supplemenation and 30 minutes after.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Maciejczyk, prof.dr, Principal Investigator — University of Physical Education, Kraków, Poland
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drwal A, Palka T, Tota L, Wiecha S, Cech P, Strzala M, Maciejczyk M. Acute effects of multi-ingredient pre-workout dietary supplement on anaerobic performance in untrained men: a randomized, crossover, single blind study. BMC Sports Sci Med Rehabil. 2024 Jun 9;16(1):128. doi: 10.1186/s13102-024-00918-1. PMID 38853269